CLINICAL TRIAL: NCT01406327
Title: Drug Use Investigation for VOLIBRIS® (Ambrisentan) (Pulmonary Arterial Hypertension)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114782
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Hypertension, Pulmonary
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — ambrisentan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects prescribed ambrisentan: Subjects with pulmonary arterial hypertension (PAH) prescribed ambrisentan during study period
  Interventions: Drug: Ambrisentan

INTERVENTIONS:
Drug: Ambrisentan — Ambrisentan

SUMMARY:
The objective of this post-marketing surveillance study is to evaluate the incidence of adverse events in Japanese subjects with pulmonary arterial hypertension treated with ambrisentan basd on prescribing information under the conditions of general clinical practice and also to grasp the following items;

1. Unknown adverse drug reactions (ADRs)
2. Incidence of ADRs to medical products in actual clinical practice
3. Factors influencing safety of ambrisentan
4. Factors influencing efficacy of ambrisentan
5. Prognosis of subjects as well as efficacy and safety of ambrisentan in long-term use (VOLIBRIS® is a trademark of Gilead Sciences, Inc,. that GSK uses under license.)

ELIGIBILITY:
Inclusion Criteria:

* Must use ambrisentan for the first time

Exclusion Criteria:

* Subjects with hypersensitivity to ambrisentan
* Subjects who is pregnant or might be pregnant
* Subjects with severe hepatic disorder

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All Japanese subjects who have received ambrisentan for the first time for the treatment of pulmonary arterial hypertension (PAH) and have given their consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2010-12-14 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
The number of adverse events in Japanese subjects with pulmonary arterial hypertension treated with ambrisentan | 1 year
The onset statuses of anemia, fluid retention, cardiac failure and hemorrhage | 1 year
The number of adverse events and clinical course in subjects with hepatic dysfunction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Takahashi T, Hayata S, Kobayashi A, Onaka Y, Ebihara T, Hara T. Surveillance on The Safety and Efficacy of Ambrisentan (Volibris Tablet 2.5 mg) in Patients with Pulmonary Arterial Hypertension in Real Clinical Practice: Post-marketing Surveillance (Interim Analysis Report). Clin Drug Investig. 2018 Mar;38(3):219-229. doi: 10.1007/s40261-017-0602-4. PMID 29282676